CLINICAL TRIAL: NCT02596321
Title: A Randomized, Double-blind, Placebo-controlled Study Investigating the Immunologic Effects and Safety of 60-day Treatment of the ALK HDM Tablets in Adult Subjects With Allergic Rhinitis and/or Atopic Asthma Induced by House Dust Mites
Brief Title: A Study Investigating the Immunologic Effects and Safety of 60-day Treatment of the ALK HDM Tablets in Adult Subjects With HDM-Induced Allergic Rhinitis and/or Atopic Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Collaborators: Linical Co., Ltd. (Industry); Datamap (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MITI3001
Record Dates: First submitted 2015-11-02; First posted 2015-11-04 (Estimated); Results first posted 2017-12-18 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Allergy; Asthma; Rhinitis
Keywords: House Dust Mite
MeSH Terms: conditions — Hypersensitivity; Asthma; Rhinitis | interventions — Allergens

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mitizax ALK HDM tablet (Experimental): Standardised allergen extract from the house dust mites Dermatophagoides pteronyssinus and Dermatophagoides farinae developmental unit, dose standard for ALK HDM tablets (12DU)
  Interventions: Drug: Mitizax
- Placebo tablet (Placebo Comparator): Placebo tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mitizax — Allergen extract
  Other Names: ALK HDM tablet; allergen extract
  Arms: Mitizax ALK HDM tablet
Drug: Placebo — Placebo tablet
  Other Names: Placebo tablet
  Arms: Placebo tablet

SUMMARY:
To demonstrate superiority of ALK HDM tablets versus placebo in immune response, measured as change of D.farinae specific immunoglobulin G4 (IgG4) from baseline to end of treatment with ALK HDM tablets given once daily over 60 days.

DETAILED DESCRIPTION:
To demonstrate superiority of ALK HDM tablets versus placebo in the immune response, measured as change of D. Farinae specific IgG4 from baseline to end of treatment with ALK HDM tablets given once daily over 60 days

To evaluate the immune response, measured as change of D. pteronyssinus, D. farinae specific immunoglobulin E (IgE) and D. pteronyssinus specific IgG4 from baseline to end of treatment with ALK HDM tablets given once daily over 60 days, compared to placebo

To evaluate in patients with HDM-allergic respiratory disease the safety and tolerability of 60-day treatment with ALK HDM tablets compared to placebo

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained before entering the study
* Patients 18-65 years of age, with a clinical history consistent with HDM-induced allergic rhinitis or allergic rhinoconjunctivitis with or without HDM-induced allergic atopic asthma for more than 1 year
* Use of symptomatic treatment of HDM-induced allergic rhinitis and/or HDM-induced atopic asthma, i.e. antihistamines, nasal decongestants, nasal and/or inhaled corticosteroid for more than 1 year
* if HDM-induced atopic asthma is present, it should be of mild to moderate severity, controlled on treatment corresponding to steps 1-3 of The Global initiative for asthma (GINA)
* Positive skin prick test response (wheal diameter ≥3 mm) to D pteronyssinus and/or D.farinae
* Moderate or higher level of D.pteronyssinus and/or D.farinae specific IgE (defined as ≥IgE Class 2; or ≥0.70 kilo unit (kU)/L)
* Patient one of the following:

  1. Male
  2. Female, infertile
  3. Female, with a negative pregnancy test and willingness to practice appropriate contraceptive methods until treatment with study drug has been discontinued.
* Patient willing and able to comply with study protocol

Exclusion Criteria:

* Previous treatment with HDM immunotherapy for more than 1 month within the last 5 years
* Ongoing treatment with any allergen-specific immunotherapy product
* Reduced lung function (defined as Forced expiratory volume in 1 second (FEV1) < 70% of predicted value after adequate pharmacologic treatment) measured at Visit 1 and Visit 2
* Clinical history of uncontrolled asthma within 3 months prior to the screening visit
* Having experienced a severe asthma exacerbation within 3 months prior to screening visit
* Symptoms of or treatment for upper respiratory tract infection, acute sinusitis, acute otitis media or other relevant infectious process at randomization
* Inflammatory conditions in the oral cavity with severe symptoms such as oral lichen planus with ulcerations or severe oral mycosis at randomization
* History of anaphylaxis with cardiorespiratory symptoms (immunotherapy, exercise-induced, food allergy, drugs or an idiopathic reaction)
* History of recurrent generalized urticaria (defined as two or more episodes) during the last 2 years
* A history of drug induced (incl. immunotherapy) facial angioedema or a family (parents and siblings) history of hereditary angioedema
* Any chronic disease (e.g. cystic fibrosis, malignancy, malabsorption or malnutrition, renal or hepatic abnormality or any other diseases that in the opinion of the investigator would interfere with the study evaluations or the safety of the subject)
* Systemic disease affecting the immune system (e.g. autoimmune disease, immune complex disease, or immune deficiency disease whether acquired or not)
* Immunosuppressive treatment (ATC code L04 or L01) within 3 months prior to the screening visit
* Currently treated with tricyclic antidepressants; catecholamine-O-methyltransferase (COMT) inhibitors and mono amine oxidase inhibitors (MAOIs) and beta-blockers including topical administration
* Use of medication at the screening visit which at the time of skin prick test (SPT) can interfere with the result (i.e. antihistamines)
* Use of an investigational drug within 30 days/5 half-lives of the drug (which ever longest) prior to the screening visit
* History of allergy, hypersensitivity or intolerance to a excipient in the investigational medicinal product (except D.Pteronyssinus and D.farinae)
* Being immediate family of the investigator or study staff, defined as the investigator's/staff's spouse, parent, child, grandparent or grandchild
* Severe mental disorders that in the opinion of the investigator would interfere with the study evaluations or the safety of the subject
* Cardiovascular conditions in which complications are possible when using adrenaline
* Women who are pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2015-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dmitri Kazei, MD, Study Director — Abbott
Locations (9):
- Belarus (2):
  - Minsk Regional Clinical Hospital, Minsk
  - City Clinical Hopsital #10, Minsk
- Russia (7):
  - Kazan State Medical Academy, Kazan'
  - National Research Center - Institute of Immunology Federal Medical-Biological Agency of Russia, Moscow
  - "Russian Medical Academy of Postgraduate Education Studies, Moscow
  - City out-patient's clinic # 94, Saint Petersburg
  - Smolensk State Medical Academy, Smolensk
  - Hospital of Russian Academy of Science, Troitsk
  - Bashkirskiy State Medical University, Ufa

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mitizax ALK HDM Tablet | Placebo Tablet
Started | 56 | 56
Completed | 53 | 56
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mitizax ALK HDM Tablet | Placebo Tablet | Total
Number analyzed (Participants) | 56 | 56 | 112
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 1 | 4
  Between 18 and 65 years | 53 | 55 | 108
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (9.1) | 31.4 (9.8) | 31.6 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 32 | 59
  Male | 29 | 24 | 53
Region of Enrollment [Count of Participants; unit: Participants]
  Belarus | 12 | 12 | 24
  Russia | 44 | 44 | 88

OUTCOME MEASURES:

1. Primary Outcome: D. Farinae Specific IgG4 Change From Baseline to End of Treatment
Description: primary efficacy endpoint of D. Farinae specific IgG4 change from baseline to end of treatment
Time Frame: 60 days from baseline
Measure: Mean (Standard Deviation); unit: mg antibody/ml
Arm/Group | Mitizax ALK HDM Tablet | Placebo Tablet
Number analyzed (Participants) | 53 | 56
mg antibody/ml | 0.473 (1.183) | -0.01 (0.067)

2. Secondary Outcome: D. Pteronyssinus Specific IgG4 Change From Baseline to End of Treatment
Description: secondary endpoint of D. pteronyssinus specific IgG4 change from baseline to end of treatment
Time Frame: 60 days from baseline
Measure: Mean (Standard Deviation); unit: mg antibody/ml
Arm/Group | Mitizax ALK HDM Tablet | Placebo Tablet
Number analyzed (Participants) | 53 | 56
mg antibody/ml | 0.455 (1.210) | 0.001 (0.076)

3. Secondary Outcome: D. Farinae Specific IgE Change From Baseline to End of Treatment
Description: the secondary endpoint of D. farinae specific IgE change from baseline to end of treatment compared to placebo
Time Frame: 60 days from baseline
Measure: Mean (Standard Deviation); unit: kUA/L
Arm/Group | Mitizax ALK HDM Tablet | Placebo Tablet
Number analyzed (Participants) | 53 | 56
kUA/L | 140.37 (288.15) | -5.56 (16.30)

4. Secondary Outcome: D. Pteronyssinus Specific IgE Change From Baseline to End of Treatment
Description: the secondary endpoint of D. pteronyssinus specific IgE change from baseline to end of treatment compared to placebo
Time Frame: 60 days from baseline
Measure: Mean (Standard Deviation); unit: kUA/L
Arm/Group | Mitizax ALK HDM Tablet | Placebo Tablet
Number analyzed (Participants) | 53 | 56
kUA/L | 124.85 (286.90) | -5.16 (27.27)

ADVERSE EVENTS:
Arm/Group | Mitizax ALK HDM Tablet | Placebo Tablet
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/56
Other Adverse Events (participants affected / at risk) | 14/56 | 4/56
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mitizax ALK HDM Tablet (N=56) | Placebo Tablet (N=56)
Oral soft tissue signs and symptoms (Gastrointestinal disorders) | 9 (9) | 1 (1)
Tongue signs and symptoms (Gastrointestinal disorders) | 3 (3) | 0 (0)
Upper respiratory tract infections (Infections and infestations) | 0 (0) | 3 (3)
Upper raspiratory tract signs and symptoms (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 0 (0)
Headaches NEC (Nervous system disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No